CLINICAL TRIAL: NCT06629571
Title: The Effect of Education Given to Patients Before Abdominal Surgery on Anxiety: A Randomized Controlled Study
Brief Title: The Effect of Preoperative Education on Anxiety
Acronym: Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MarmaraU Banu Gümüş01
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Surgery; Anxiety
Keywords: SurgeryAnxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patient education
  Interventions: Other: Education
- Control (No Intervention): No patient education

INTERVENTIONS:
Other: Education — Training for the patient before surgery
  Other Names: Surgery Education
  Arms: Experimental

SUMMARY:
This randomized controlled study aimed to evaluate the effect of preoperative education on anxiety levels in patients undergoing abdominal surgery at a training hospital in Istanbul. The study population included patients admitted between January and June 2024. After power analysis, patients were divided into experimental (n=40) and control (n=41) groups. The experimental group received preoperative information, while the control group received standard care. Anxiety levels were assessed using the State-Trait Anxiety Inventory (STAI). Data were analyzed with SPSS, using tests such as the Mann-Whitney U and Wilcoxon Sign tests.

DETAILED DESCRIPTION:
As a result of this study, the anxiety levels of patients who received preoperative information training in the prevention or reduction of anxiety were found to be lower than patients who received routine care. The lower score indicated that they experienced less anxiety or were able to manage their anxiety in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the general surgery clinic for abdominal surgery in category A-B-C
* must be over the age of 18
* To be literate- to be a writer
* Being conscious
* Who does not have a psychiatric disorder

Exclusion Criteria:

* Exit the research during the study,
* Group D and E abdominal surgery has been performed
* don't be under the age of 18
* Unconscious patient,
* Who has a psychiatric disorder
* Patients with communication disabilities or who cannot speak Turkish were determined as patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
STAI Form TX I,STAI Form TX II | 1 Day before the operation and 1 day after the operation
  In the scoring of both scales, the total score of reversed statements is subtracted from the total score obtained from direct statements, and 50 points are added as a fixed value for STAI TX-I and 35 points for STAI TX-II. The score obtained as a result of this calculation is the individual's anxiety score. The scores obtained from both scales theoretically vary between 20 and 80. A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety. The STAI TX-I threshold is 39-40 points. Mild anxiety is between 20-31 points, moderate anxiety is between 32-42 points, and anxiety is above 42-44 points. Since it shows how the person feels at that moment, regardless of the situation and conditions they are in, the threshold is accepted as 44-45 points in patients in the pre-operative period. A score between 40-59 points is considered moderate, and a score between 60-80 points is considered high.

CONTACTS AND LOCATIONS:
Locations (1):
- MarmaraU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No